CLINICAL TRIAL: NCT04013997
Title: Safety of Exoskeleton-assisted Walking in SCI Inpatient Rehabilitation
Brief Title: Exoskeleton-assisted Walking in SCI Inpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Miguel Escalon, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: GCO 15-2253
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries; Inpatients
Keywords: Rehabilitation; Walking; Equipment and Supplies
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Prospective subjects were recruited following admission to the SCI inpatient unit at Mount Sinai Hospital. Attending physicians and rehabilitation clinicians identified patients admitted to the unit who may be eligible for the study. Consent forms were given to prospected participants. After enrolling into the study, participants received locomotor training with the exoskeleton as part of their acute inpatient rehabilitation using the Ekso. Standing and walking with the Ekso started as soon as the clinical team determined it was safe for participants to begin standing, and continued until the participant was discharged from inpatient rehabilitation. The study team monitored participants for adverse events (safety), tracked the amount of walking provided during the inpatient stay (feasibility), and explored the improvement of activities of daily living compared to matched control group who didn't have Ekso training chosen from retrospective chart review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Exoskeletal-assisted walking training group (Experimental): Prospective subjects were recruited following admission to the SCI inpatient unit at Mount Sinai Hospital. Attending physicians and rehabilitation clinicians identified patients admitted to the unit who may be eligible for the study.
  Interventions: Device: EksoGT
- Matched control group (No Intervention): Twenty inpatients with SCI were identified as the matched control group through reviewing an acute inpatient rehabilitation database of Uniform Data System for Medical Rehabilitation by a person blinded to the study.
  The control group received a minimum of 15 hours of standard of care, including physical and occupational therapy, for acute inpatient rehabilitation per week. The control groups received the same amount of acute rehabilitation time per week as the intervention group.

INTERVENTIONS:
Device: EksoGT — The intervention group received a minimum of 15 hours of standard of care, including physical and occupational therapy, for acute inpatient rehabilitation per week. After enrolling into the study, participants received locomotor training with the exoskeleton as part of their acute inpatient rehabilitation using the Ekso. Standing and walking with the Ekso started as soon as the clinical team determined it was safe for participants to begin standing, and continued until the participant was discharged from inpatient rehabilitation.
  Other Names: Exoskeletal-assisted walking training
  Arms: Exoskeletal-assisted walking training group

SUMMARY:
To assess how safe the exoskeleton, EksoGT, is to use for acute inpatient rehabilitation, if it helps people to walk better than with traditional walking training methods, or if they have any other effects (better or worse) on recovery.

DETAILED DESCRIPTION:
Wearable robots that assist with walking over ground are now available in rehabilitation centers. However, the study team did not know how soon it is safe to start using these devices for rehabilitation, if they helped people to walk better than with traditional locomotor training methods, or if they had any other effects (better or worse) on recovery.

The study team's objectives of this study were to explore the safety, feasibility, and efficacy of using the powered exoskeleton, EksoGT, to provide a locomotor training intervention in acute inpatient rehabilitation for persons with spinal cord injury (SCI) who were eligible for locomotor training.

Aim 1 examined the safety of exoskeleton use for persons with SCI during inpatient rehabilitation. Measures for this aim analyzed the amount of falls as well as types and counts of other adverse events (AE) for both serious and non-serious events as outlined by the FDA.

Aim 2 helped determine the feasibility of exoskeleton use during inpatient rehabilitation for SCI by monitoring the time from admission to first stand in the device, accumulated step count/time in the device, and progression of locomotor training frequency, duration, and intensity.

Aim 3 explored the potential for associations between exoskeleton use in inpatient rehabilitation and body functions and activities associated with walking. Measures for this aim included: American Spinal Injury Association (ASIA) Impairment Scale (AIS), Neurological Level of Injury (NLI), Upper and Lower Extremity Motor Scores, and Functional Index Measure (FIM).

Prospective subjects were recruited following admission to the SCI inpatient unit at Mount Sinai Hospital. Attending physicians and rehabilitation clinicians would identify patients admitted to the unit who may be eligible for the study. Consent forms were given to prospected participants.

After enrolling into the study, participants received locomotor training with the exoskeleton as part of their acute inpatient rehabilitation using the Ekso. Standing and walking with the Ekso started as soon as the clinical team determines it is safe for participants to begin standing, and continued until the participant is discharged from inpatient rehabilitation. The study team monitored participants for adverse events (safety), tracked the amount of walking provided during the inpatient stay (feasibility), and explored the improvement of activities of daily living (functioning) compared to the matched control group who didn't have Ekso training and were chosen by a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Height between 5'2" and 6'2" (1.6 meters to 1.9 meters)
* Weight less than 220 pounds (100 kilograms)
* Near Normal range of motion (ROM), as follows:
* Hip: 5 degrees of extension; 110 of flexion
* Knee: Full extension to 110 of flexion
* Ankle: at least 0 of dorsiflexion to 25 of plantarflexion
* Are eligible for locomotor training as part of inpatient rehabilitation
* Independent with static sitting balance
* Sufficient function upper extremity strength to manage walking aid (front-wheeled walker, platform walker, or crutches)
* Able to follow directions

Exclusion Criteria:

* Uncontrolled cardiovascular conditions (i.e. heart failure, angina, hypertension)
* Inability to stand upright due to orthostatic hypotension
* Body characteristics that do not fit within exoskeleton limits
* Upper leg length discrepancy > 0.5" or lower leg discrepancy >0.75"
* Skin integrity issues in areas that would contact the device or that would likely be made worse by device use
* Pregnancy
* Colostomy
* Non-English Speaking
* The participant is able to walk better with exoskeleton assistance at baseline
* Any other issue that might prevent safe standing or walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of fall | 2 years
  Number of falls to assess safety
Number of adverse events | 2 years
  types and counts of the adverse events for both serious and non-serious events as outlined by the FDA to assess safety

SECONDARY OUTCOMES:
The time from admission to first stand in the device | 2 years
  The days between admission date and the date of first stand in the device
Accumulated step count in the device | 2 years
  The total steps count during the exoskeletal-assisted walking (EAW) training in the acute inpatient rehabilitation
Accumulated step time in the device | 2 years
  The total walking time during the EAW training in the acute inpatient rehabilitation
Proportion of walking time | 2 years
  The change of the proportion of walking time in the device (proportion of walking time = walking time/total time in the device)
American Spinal Injury Association (ASIA) Impairment Scale (AIS) | 2 years
  A: Complete - No motor or sensory function is preserved in the sacral segments S4-S5.
  B: Incomplete - Sensory function preserved but not motor function is preserved below the neurological level and includes the sacral segments S4-S5.
  C: Incomplete - Motor function is preserved below the neurological level, and more than half of key muscles below the neurological level have a muscle grade less than 3.
  D: Incomplete - Motor function is preserved below the neurological level, and at least half of key muscles below the neurological level have a muscle grade of 3 or more.
  E: Normal - Motor and sensory function are normal.
Neurological Level of Injury (NLI) | 2 years
  The NLI refers to the most caudal segment of the spinal cord with normal sensory and antigravity motor function on both sides of the body
Upper Extremity Motor Scores (UEMS) | 2 years
  Total score from 0-50, with higher score indicating better outcomes
Lower Extremity Motor Scores (LEMS) | 2 years
  Total score from 0-50, with higher score indicating better outcomes
Functional Independence Measure (FIM) | 2 years
  The FIM is an 18-item instrument, total score range from 18-126, with higher score indicating higher level of function

CONTACTS AND LOCATIONS:
Overall Officials: Miguel X Escalon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No